CLINICAL TRIAL: NCT01023880
Title: An Open-Label Study to Determine the Maximum Tolerated Dose and Evaluate the Efficacy and Safety of CEP-18770 in Patients With Relapsed Multiple Myeloma Refractory to the Most Recent Therapy
Brief Title: Study to Determine the Maximum Tolerated Dose and Evaluate the Efficacy and Safety of CEP-18770 (Delanzomib) in Patients With Relapsed Multiple Myeloma Refractory to the Most Recent Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18770/2043
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — delanzomib

ARMS (1):
- 1 (Experimental): CEP-18770
  Interventions: Drug: CEP-18770

INTERVENTIONS:
Drug: CEP-18770 — CEP-18770 beginning at a dose of 1.5 mg/m2. Patients will receive I.V. administration on days 1, 8, 15 (up to 8 cycles of 28 days each). When the MTD is established, additional patients will be treated at the MTD.
  Other Names: delanzomib

SUMMARY:
The primary objective for part 1 of the study is to determine the maximum tolerated dose (MTD) of CEP-18770 in patients with relapsed and refractory multiple myeloma. The primary objective for part 2 is to evaluate the antitumor activity of CEP-18770 in patients treated at the MTD.

ELIGIBILITY:
Key Inclusion Criteria:

The patient has:

* relapsed multiple myeloma that has progressed following therapies that included bortezomib and an IMiD (thalidomide or lenalidomide) either alone or in any combination.
* multiple myeloma, which is refractory to the most recent therapy (bortezomib or IMiD, or any other chemotherapy), or the patient did not tolerate and discontinued the most recent therapy for multiple myeloma but has recovered from its toxic effects.
* measurable disease defined as 1 of the following:

  * serum M-protein ≥0.5 g/dL
  * urine M-protein ≥200 mg/24 hours
* a life expectancy of more than 3 months.
* an ECOG performance status of 0, 1, or 2.
* adequate hepatic organ function.
* an absolute neutrophil count (ANC), hemoglobin level, and platelet count within protocol-specific ranges.
* been independent of granulocyte-colony stimulating factor (G-CSF) or granulocyte macrophage-colony stimulating factor (GM-CSF) support for more than 1 week.
* been independent of platelet transfusion for more than 1 week.
* received, or may have received, an allogeneic and/or autologous transplant.
* a creatinine clearance of 30 mL/minute or more as measured or as calculated based on the Cockcroft-Gault method.
* if the patient is a female of childbearing potential (not surgically sterile or 1 year postmenopausal): must use a medically accepted method of contraception (including abstinence) and must agree to continue use of this method for the duration of the study and for 3 months after participation in the study.
* if the patient is a male: is surgically sterile, or if sexually active, is currently using an effective barrier method of contraception, and agrees to continue use of this method for the duration of the study and for 3 months after the last administration of study drug.

Key Exclusion Criteria:

The patient:

* has nonmeasurable multiple myeloma.
* received glucocorticoid therapy (prednisone >10 mg/day orally or equivalent) within the last 2 weeks prior to the first dose of study drug.
* has POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy or monoclonal proliferative disorder, and skin changes).
* has plasma cell leukemia.
* received chemotherapy with approved anticancer therapeutics within 2 weeks, or within 5 drug half-lives (t1/2), or investigative anticancer therapeutics within 4 weeks, or within 5 drug half-lives (t1/2), before the first dose of study drug, whichever time is greater.
* received radiation therapy or immunotherapy in the 4 weeks prior to, or localized radiation therapy within 1 week prior to, the first dose of study drug.
* received prior treatment with CEP-18770.
* has used a medication known to be a potent inducer of CYP2E1, CYP2D6 or CYP3A4/5 within 4 weeks prior to the first dose of study drug.
* has used a medication known to be a potent inhibitor of CYP2E1, CYP2D6 or CYP3A4/5 within 2 weeks prior to the first dose of study drug.
* had major surgery within 3 weeks before the first dose of study drug.
* has congestive heart failure or had symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within the last 6 months.
* had an acute infection requiring systemic antibiotics, antiviral agents, or antifungal agents within 2 weeks before the first dose of study drug.
* has a known or suspected human immunodeficiency virus (HIV) infection on the basis of medical history.
* had a nonhematologic malignancy within the past 3 years except for the following: adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or breast, or prostate cancer (Gleason grade <6 with prostate specific antigen (PSA) levels within the normal range).
* has myelodysplastic or myeloproliferative syndrome.
* has significant neuropathy.
* is a pregnant or lactating woman. Any women becoming pregnant during the study will be withdrawn from the study.
* has known central nervous system involvement.
* has any serious psychiatric or medical condition that could interfere with treatment or study procedures, place the patient at unacceptable risk, or hinder the interpretation of study data.
* has known hypersensitivity to mannitol or hydroxypropyl betadex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Every 4 weeks, until completion of treatment

SECONDARY OUTCOMES:
Elapsed time from the ORR date to the date of disease progression (DOR) | at disease progression
Elapsed time from the date of first dose of CEP-18770 to the date of first response (TTR) to treatment with CEP-18770 | at date of first response (TTR) to treatment
Elapsed time from the date of first dose of CEP-18770 to the date of disease progression (TTP) | at date of disease progression (TTP)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (13):
- United States (13):
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford Heme Group, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Northwestern University Medical School, Chicago, Illinois
  - Henry Ford Health System Protocol Review Committee, Detroit, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Vogl DT, Martin TG, Vij R, Hari P, Mikhael JR, Siegel D, Wu KL, Delforge M, Gasparetto C. Phase I/II study of the novel proteasome inhibitor delanzomib (CEP-18770) for relapsed and refractory multiple myeloma. Leuk Lymphoma. 2017 Aug;58(8):1872-1879. doi: 10.1080/10428194.2016.1263842. Epub 2017 Jan 31. PMID 28140719